CLINICAL TRIAL: NCT06019741
Title: Rivaroxaban and Aspirin Versus Aspirin Alone in Preventing Atherothrombotic Events in Patients Following Coronary Artery Bypass Graft Surgery
Brief Title: Rivaroxaban Post Coronary Bypass Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shiraz University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Javad Kojuri, professor, Shiraz University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IR.SUMS.MED.REC.1401.411
Record Dates: First submitted 2023-08-25; First posted 2023-08-31 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Post Coronary Bypass Surgery Patients
Keywords: coronary bypass surgery; aspirin; rivaroxaban; MACE
MeSH Terms: interventions — Rivaroxaban

STUDY DESIGN:
Intervention Model Description: randomized double blind of placebo and intervention group
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: simple randomization
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- aspirin and rivaroxaban (Experimental): post coronary bypass patients, received aspirin 80 mg and rivaroxaban 2.5 mg PO twice daily
  Interventions: Drug: Rivaroxaban and aspirin 80
- aspirin (Active Comparator): post coronary bypass patients, received aspirin 80 mg
  Interventions: Drug: Aspirin 80

INTERVENTIONS:
Drug: Rivaroxaban and aspirin 80 — rivaroxaban 2.5 mg twice daily orally added to aspirin 80 mg post coronary bypass surgery
  Arms: aspirin and rivaroxaban
Drug: Aspirin 80 — aspirin 80 mg orally post coronary bypass surgery
  Arms: aspirin

SUMMARY:
Post coronary bypass patients were randomized to receiving aspirin alone or aspirin and low dose rivaroxaban

DETAILED DESCRIPTION:
This study is a 1-year randomized, double-blind placebo-controlled trial to evaluate the effects of adding rivaroxaban to the treatment of patients after coronary bypass surgery. All patients referred for either off-pump or on-pump coronary bypass surgery to 3 academic hospitals in Shiraz, Iran were screened according to inclusion criteria. Clinicians at these sites were informed of this study and asked to refer patients after coronary bypass surgery.

A total of 414 patients were initially included in the study, but 171 of them were excluded based on the exclusion criteria (Figure 1). The remaining 243 patients were then randomly divided into two groups: group 1, receiving aspirin 80 mg daily plus placebo; group 2, receiving aspirin 80 mg daily plus rivaroxaban 2.5 mg twice daily.

Clinical outcomes were assessed at the end of first year post-operation. Subjects will undergo a complete history and physical examination and the study variables were assessed. Patients were followed every 2 weeks for any occurrence at these visits, patients' compliance was assessed, standard medication was adjusted as appropriate, and all interventions, outcome events, and adverse events were recorded. The patients were followed for the occurrence of major adverse cardiac events (MACE), defined as follows: 1) cardiogenic death; 2) myocardial infarction (hospital visit for myocardial infarction reported by patient or hospital admission for myocardial infarction reported by cardiologist); and 3) cerebrovascular accidents. Occurrence of major bleeding and chest pain, and functional capacity exercise (assessed with exercise tolerance test) were also evaluated. Additional variables that will be collected at baseline include demographic and clinical characteristics of patients as follows: sex (male, female), age (mean (SD)), hypertension (yes/no), and diabetes mellitus (yes/no).

To document any unfavorable occurrences, the patients were questioned via telephone monthly about any potential side effects.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 undergoing primary isolated coronary bypass surgery, with or without cardiopulmonary bypass

Exclusion Criteria:

* Other cardiac surgeries except for coronary bypass surgery
* Left ventricular ejection fraction < 30 %
* Liver disease
* Clopidogrel or aspirin intake within 7 days of operation
* Need for perioperative warfarin
* Active gastroduodenal ulcer or post-operative gastrointestinal bleeding
* Profuse post-operative pleural effusion (drainage >200 ml/h for 2 h or more
* Postoperative low cardiac output syndrome or requirement for high levels of hemodynamic support (more than 2 inotropes for more than 24 h and/or intra-aortic balloon pump)
* Clinical instability, such as perioperative myocardial infarction or malignant tumor.

Ages: 45 Years to 87 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-07-20 (Actual)

PRIMARY OUTCOMES:
MACE | 1 year
  Major adverse cardiac events (MACE), defined as follows: 1) cardiogenic death; 2) myocardial infarction (hospital visit for myocardial infarction reported by patient or hospital admission for myocardial infarction reported by cardiologist) ,and 3) cerebrovascular accidents
bleeding | 1 year
  all types of reported bleeding, major or minor

SECONDARY OUTCOMES:
functional capacity | 1 year
  functional capacity assessed by exercise tolerance test, based on METS, duration of toleration of exercise

CONTACTS AND LOCATIONS:
Locations (1):
- Professor Kojuri Cardiology Clinic, Shiraz, Fars, Iran

IPD SHARING:
Plan to Share IPD: No
Data is available in professor kojuri registry, and will be available upon rational request